CLINICAL TRIAL: NCT02929238
Title: Polypropylene Suture Interfaced Between Wound and Negative Pressure Wound Therapy to Reduce Pain: a Pilot Study
Brief Title: Wound Vac Polypropylene Suture Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: pro00049555
Record Dates: First submitted 2016-10-07; First posted 2016-10-11 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Wound Vac; Suture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polypropylene Suture Right Side (Experimental): Polypropylene suture will be placed over half the wound. There is an equal chance for the suture to be placed on the right or left through randomization. THe other half of the wound will not have the suture placed on it and will act as the control. The wound vac will be placed over entire wound.
  Interventions: Other: Polypropylene Suture Right Side
- Polypropylene Suture Left Side (Experimental): Polypropylene suture will be placed over half the wound. There is an equal chance for the suture to be placed on the right or left through randomization. THe other half of the wound will not have the suture placed on it and will act as the control. The wound vac will be placed over entire wound.
  Interventions: Other: Polypropylene Suture Left Side

INTERVENTIONS:
Other: Polypropylene Suture Right Side — Suture Description: The suture used in this study will be a sterilized polypropylene suture and individually crossed in the base of the wound. Polypropylene is commonly used for commercially available implanted meshes. The polypropylene suture is intended for single use only and the individual suture will be packaged and purchased sterile.
  Arms: Polypropylene Suture Right Side
Other: Polypropylene Suture Left Side — Suture Description: The suture used in this study will be a sterilized polypropylene suture and individually crossed in the base of the wound. Polypropylene is commonly used for commercially available implanted meshes. The polypropylene suture is intended for single use only and the individual suture will be packaged and purchased sterile.
  Arms: Polypropylene Suture Left Side

SUMMARY:
You are being asked to participate in this study because you have a complex wound that requires treatment with negative pressure wound therapy (NPWT). NPWT is a therapeutic technique which involves the placement of a wound vacuum at the site of the wound. The wound vacuum delivers a negative pressure at the wound site through a dressing. Any fluid collected during this process is collected through a foam (sponge) underneath the dressing. This therapy helps to draw the edges of the wound together, while removing infectious material, to help promote healthy tissue growth and speed up wound healing. The purpose of this study is to determine if placing polypropylene suture (a material normally used to close wounds) between the wound and the NPWT foam would decrease pain upon removal of the sponge while allowing adequate healing of the wound.

DETAILED DESCRIPTION:
If you decide to participate in the study you will be asked to sign this informed consent form prior to beginning any study activities. If you agree to participate the study procedures are as follows:

* The participants enrolled in this study will receive NPWT in combination with polypropylene suture being laid out over half of the wound. Enrollment in this study is not considered standard of care.

  * You will be randomized (like flipping a coin) to what side of the wound the suture will be placed on. Randomization means the study team has no say in what side the suture goes on. Your information is put into a computer and the computer picks what side to place the suture. The polypropylene suture will be placed over half of your wound. There is an equal chance for the polypropylene suture to be placed on the right or left side. The other half of your wound will not have the polypropylene suture in place and will act as the control (comparison) group in this study. The use of the study polypropylene suture is not considered standard of care.
* The wound vacuum will be placed over the entire wound and will be left in place for no more than 3 days as per standard of care.
* After no more than 3 days at a time during the healing process, the nurses will remove the wound vacuum, dressings, suture, and the sponge.
* One blinded (they are not told which side of the wound the suture is placed on) study physician will come look at your wound. This study physicians will determine if further NPWT, with or without the study polypropylene suture, is needed.
* You will be asked to complete a pain rating questionnaire (rating scale 0-10) in relation to both sides of your wound when the wound vacuum has been removed.
* If further NPWT is needed without the use of the study polypropylene suture, you will be withdrawn from the study
* If discharged with NPWT you will not continue receive polypropylene suture placement and that would be end of study participation
* If further NPWT is needed with the use of negative pressure wound therapy, the polypropylene suture and the sponge will be placed and the process will continue as noted above until your wound is healed or you are withdrawn from the study.
* Information from your medical records will be collected throughout this study. You will also be asked questions about your medical and surgical history as well as what medications you are currently taking.
* Your demographics will be collected including your age, date of birth, race, sex, height, weight, and ethnicity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 years or older
2. All patients with an open wound who require NPWT
3. Hospitalized patient in need of NPWT for ≥ 6 days
4. Willingness to comply with protocol, complete study assessments (pain scale ratings), allow pictures to be taken, and provide written informed consent

Exclusion Criteria:

1. Male or female less than 18 years of age
2. Prisoners
3. Outpatients
4. Patients with infected wounds
5. Patients with poor blood flow
6. Hospitalized patient in need of NPWT for < 6 days
7. Not willing to provide written informed consent or remain in compliance with the study protocol requirements

Prisoners will be excluded from this study as they are considered an at risk population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-06; Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
Pain Rating Questionnaire | no longer than 6 months
  testing to see if suture decreases the pain when removing the wound vac

SECONDARY OUTCOMES:
Blinded Physician Interpretation | no longer than 6 months
  one blinded physician looks at wound to make sure the suture is not interfering with wound healing

CONTACTS AND LOCATIONS:
Overall Officials: John Cull, M.D., Principal Investigator — Prisma Health-Upstate
Locations (1):
- Greenville Health System, Greenville, South Carolina, United States